CLINICAL TRIAL: NCT01861405
Title: Neurocognitive and fMRI Activation Changes Observed at Baseline and After Whole Brain Radiation vs. Radiosurgery for Patients With Cerebral Metastases: a Prospective Case-control Analysis.
Brief Title: Neurococognitive and Functioal Assessment of Patients With Brain Metastases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Other Study IDs: 13D.02
Record Dates: First submitted 2013-05-20; First posted 2013-05-23 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Cerebral Metastases Patients
MeSH Terms: interventions — Neuropsychological Tests; Spermine Synthase; Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Cerebral metastases subjects: Prior to each subject's radiation treatment (either whole brain radiation therapy or stereotactic radiosurgery), he/she will have fMRI scanning and neuropsychological testing and conduct a quality of life assessment. Each subject will then have standard of care WBRT or SRS treatment. Following WBRT or SRS treatment, subjects will have 4 month follow up fMRI scanning, and have neuropsychological testing and a quality of life assessment 4 months and 12 months post treatment.
  Interventions: Behavioral: neuropsychological testing and quality of life assessments; Radiation: Standard of Care WBRT or SRS; Device: Functional magnetic resonance imaging
- Healthy participants: Healthy control subjects will be matched by age, gender, education, ect. to cerebral metastases subjects. Each will have fMRI scannings (3 total), neuropsychological testings (3 total), and quality of life assessments (3 total) at the same time points as their matched cerebral metastases subject.
  Interventions: Behavioral: neuropsychological testing and quality of life assessments; Device: Functional magnetic resonance imaging

INTERVENTIONS:
Behavioral: neuropsychological testing and quality of life assessments
Radiation: Standard of Care WBRT or SRS
  Groups: Cerebral metastases subjects
Device: Functional magnetic resonance imaging

SUMMARY:
The investigators seek to perform an observational study in patients with brain metastases that are to undergo whole brain radiation therapy (WBRT) or stereotactic radiosurgery (SRS) treatment in order to quantify any baseline neurocognitive changes which may result from intracranial disease burden, from radiation treatment (WBRT or SRS), or both. To do so, the investigators will compare matched control subjects to patients at time points obtained before and after radiation treatment with either SRS or WBRT. Pre-treatment evaluation will include neurocognitive testing and an assessment of fMRI task-related activation patterns and resting state brain activity. Four and twelve month post-treatment neuropsychological evaluations will be performed and pre- and 4-month post-treatment fMRI scans will be obtained in order to evaluate changes in neurocognitive functioning with a focus on short-term memory and executive function domains. A brief quality of life assessment will also be completed at each study time point. In order to plan treatment strategies in the future it is important to accurately document the effects of intracranial disease burden as well as radiation treatment on neurocognitive functioning, validate fMRI activation tasks for short term memory and executive functioning, and quantify the activation volumes that would potentially be spared in future "cognitive sparing" protocols.

The investigators hypothesize first that the amount and location of intracranial disease burden will represent pre-treatment variables that affect NCF. The compromised NCF will be visualized in both the resting state and task-oriented neurocognitive exercise. The investigators anticipate that any perturbation in resting state caused by intracranial disease burden should be reflected in patients when compared to matched controls.

The investigators hypothesize additionally that cancer patients with brain metastases undergoing radiation treatments will have improved intracranial disease control at the expense of executive and memory function with differences between patients that undergo stereotactic radiosurgery or whole brain radiation alone.

DETAILED DESCRIPTION:
This research protocol is designed to perform neuropsychological testing and fMRI scanning in patients with brain metastases that are to undergo either WBRT or SRS treatment at Thomas Jefferson University Hospital. Eligible patients will be referred through the department of Neurosurgery and Radiation-oncology. The patients will complete the informed consent for both the pre- and post-treatment (4 month after WBRT or SRS is completed) fMRI scanning and pre- and post-treatment (4 and 12 months after WBRT or SRS is completed) neuropsychological testing sessions and be told that participation in either the fMRI scans and the neuropsychological testing is voluntary. Patients will also be told that the data will be collected for observational research purposes only and will not directly affect their clinical care. Patients and their insurers will not be additionally billed as a consequence of this study aside from the clinical billing that is consistent with current clinical practice.

The fMRI study will be added on to the pre-existing treatment planning and follow up MRI scan that would be obtained out of clinical necessity without the study.

In order to be able to identify and distinguish normal versus abnormal brain activity patterns associated with the various fMRI tasks and resting state imaging procedures that are part of this study, it will be necessary to scan a subset of healthy (age, education, gender matched) normal controls on the various cognitive and behavioral tasks. This is the only way to determine the validity of the tasks used in terms of their activation properties and the normal brain areas involved in the task. Specifically, the healthy age matched controls are critical for this study as there is no other way to validate the fMRI findings with the hippocampal and executive function activations tasks. Normal matched controls are needed for proper analysis of both the neurocognitive and the neuroimaging data. For the neurocognitive data, the normal control data are needed to construct the Reliable Change Index (RCI) referenced below in the Statistics Section. Also, a comparison to normal is important for estimating the magnitude of any change observed in the patients, to determine if it has clinical relevance. For the neuroimaging data, the normal controls are needed to provide a reference or comparison point to quantify the degree to which the brain-imaging map (referred to as a Statistical Parametric Map, SPM) at each point in time (baseline, post-treatment) deviates from normal. By comparing the patient groups to normals, fMRI activation related to ancillary or idiosyncratic factors during the scan cancel out, leaving only the activation directly related to the cognitive task. Also, determining the presence of new, atypical brain activation sites, lost activation sites, or deactivations, can only be achieved by have a normal SPM brain map for comparison. This applies equally for the task-driven fMRI and the resting state functional connectivity data.

To analyze within-subject analyses with the neuroimaging data, we will examine the neuroimaging data on a within-subject but that will not be the primary quantitative approach to the imaging data, as such within-subject comparisons can be prone to methodologic problems. There is a phenomenon known in the neuroimaging literature as "double dipping" which concerns the ability to distinguish real versus random variation over time. Double dipping refers to the use of test findings at one point in time to constrain or bias the data outcomes and changes registered at a second point in time. More concretely, differences seen in the imaging data may reflect changes in the error, artifactual activations, not change in true-task related activation. To avoid this problem we operationalize change by comparing each patient's imaging data with an index of their deviation from healthy normals at each point in time (pre-surgery/baseline, and post-surgery). This procedure provides a systematic means of quantifying and then comparing the typicality of both pre and postsurgical neurocognitive activations and network organization, a procedure that alleviates concern about "double dipping". This "double dipping" phenomenon and the remedy we propose applies equally for the task-driven fMRI, the resting state functional connectivity data, and the DTI data.

In essence, the methodology proposed minimizes reliance on random, session-specific fluctuations as part of the reference or comparison point for determining change. Our method quantifies the deviation of our patients from normal, examining the relative difference in those deviations as our index of change. In so doing, we avoid the use of our pre-treatment neuroimaging results as the template for comparing and determining change, minimizing concerns of double dipping.

There is no risk associated with the scanning procedure so long as there is no metal in the body. The study of normal volunteers also allows for determination of the stability of the activation findings over time; this allows for verification of the reliability of the fMRI tasks and other procedures over time. Without an understanding of the potential normal change that can occur in brain activation and structure over time, it is impossible to determine if a pathologic change has occurred. This group of normal subjects will be studied in advance in order to validate the fMRI tasks. Furthermore, normal control subjects will be yoked or linked to matched patients and return for additional scanning sessions at the same time points as their matched patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a cumulative intracranial disease burden of up to but not exceeding 8cc.
* Patients with newly diagnosed brain metastases are undergoing WBRT or SRS as previously determined by their oncologist and or radiation oncologist.
* Right or left hand dominance.
* Karnofsky performance status (KPS) equal to or greater than 70.
* 70 years old or younger.
* All non-hematopoietic histologies except melanoma and renal cell carcinoma.
* Brainstem lesions are acceptable.
* Normal renal function to tolerate a contrast enhanced MRI scan.
* Patients must provide study specific informed consent prior to study entry.

Exclusion Criteria:

* Age less than 18 years old.
* KPS <70.
* Pregnant female.
* Active systemic disease.
* Age greater than 70 years old.
* Patients with leptomeningeal metastases.
* Contraindication for MRI such as implanted metal devices, foreign bodies or severe claustrophobia or axial back pain precluding a prolonged MRI study.
* Prior radiation therapy to the brain.
* Poor renal function rendering contrast enhanced MRI un-obtainable.
* Histological diagnosis of small cell lung cancer.
* Craniotomy or other major surgery within 2 weeks of start of either SRS or WBRT.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with brain metastases will be referred through the department of Neurosurgery and Radiation-oncology at Thomas Jefferson University Hospital. Healthy subjects will recruited through postings distributed around the hospital and university bulletin boards and through an advertisement in a local newspaper.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2013-03; Primary Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
To establish, through neurocognitive testing and fMRI, a correlation between baseline resting state functional brain connectivity, fMRI task related activation patterns and neurocognitive functioning (NCF) in patients with brain metastases. | Continuous throughout 24 month study participation

SECONDARY OUTCOMES:
To establish from normal control data a reliable change index (RCI) in order to establish the significance and magnitude of any baseline deviations in neurocognitive functioning (NCF) in patients with brain metastases. | Continuous throughout 24 month study participation
To establish through paired comparisons any significant changes from baseline in NCF and fMRI data after radiation treatmentin patients with brain metastases, adjusted respectively from a reliable change index and statistical parameters. | Continuous throughout 24 month study participation.
To utilize the data from Aims 1-3 to design a prospective randomized comparison of patient outcomes after SRS alone vs. WBRT, stratified by good and poor baseline NCF groups. | Continuous throughout 24 month study participation

CONTACTS AND LOCATIONS:
Overall Officials: Yaron Moshel, MD, PhD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Andrews DW, Scott CB, Sperduto PW, Flanders AE, Gaspar LE, Schell MC, Werner-Wasik M, Demas W, Ryu J, Bahary JP, Souhami L, Rotman M, Mehta MP, Curran WJ Jr. Whole brain radiation therapy with or without stereotactic radiosurgery boost for patients with one to three brain metastases: phase III results of the RTOG 9508 randomised trial. Lancet. 2004 May 22;363(9422):1665-72. doi: 10.1016/S0140-6736(04)16250-8. PMID 15158627
- [Background] Patchell RA, Tibbs PA, Walsh JW, Dempsey RJ, Maruyama Y, Kryscio RJ, Markesbery WR, Macdonald JS, Young B. A randomized trial of surgery in the treatment of single metastases to the brain. N Engl J Med. 1990 Feb 22;322(8):494-500. doi: 10.1056/NEJM199002223220802. PMID 2405271
- [Background] Herman MA, Tremont-Lukats I, Meyers CA, Trask DD, Froseth C, Renschler MF, Mehta MP. Neurocognitive and functional assessment of patients with brain metastases: a pilot study. Am J Clin Oncol. 2003 Jun;26(3):273-9. doi: 10.1097/01.COC.0000020585.85901.7C. PMID 12796600
- [Background] Meyers CA, Smith JA, Bezjak A, Mehta MP, Liebmann J, Illidge T, Kunkler I, Caudrelier JM, Eisenberg PD, Meerwaldt J, Siemers R, Carrie C, Gaspar LE, Curran W, Phan SC, Miller RA, Renschler MF. Neurocognitive function and progression in patients with brain metastases treated with whole-brain radiation and motexafin gadolinium: results of a randomized phase III trial. J Clin Oncol. 2004 Jan 1;22(1):157-65. doi: 10.1200/JCO.2004.05.128. PMID 14701778
- [Background] Aoyama H, Shirato H, Tago M, Nakagawa K, Toyoda T, Hatano K, Kenjyo M, Oya N, Hirota S, Shioura H, Kunieda E, Inomata T, Hayakawa K, Katoh N, Kobashi G. Stereotactic radiosurgery plus whole-brain radiation therapy vs stereotactic radiosurgery alone for treatment of brain metastases: a randomized controlled trial. JAMA. 2006 Jun 7;295(21):2483-91. doi: 10.1001/jama.295.21.2483. PMID 16757720
- [Background] Chang EL, Wefel JS, Hess KR, Allen PK, Lang FF, Kornguth DG, Arbuckle RB, Swint JM, Shiu AS, Maor MH, Meyers CA. Neurocognition in patients with brain metastases treated with radiosurgery or radiosurgery plus whole-brain irradiation: a randomised controlled trial. Lancet Oncol. 2009 Nov;10(11):1037-44. doi: 10.1016/S1470-2045(09)70263-3. Epub 2009 Oct 2. PMID 19801201
- [Background] Brem S, Panattil JG. An era of rapid advancement: diagnosis and treatment of metastatic brain cancer. Neurosurgery. 2005 Nov;57(5 Suppl):S5-9; discusssion S1-4. doi: 10.1093/neurosurgery/57.suppl_5.s4-5. PMID 16237289
- [Background] Gavrilovic IT, Posner JB. Brain metastases: epidemiology and pathophysiology. J Neurooncol. 2005 Oct;75(1):5-14. doi: 10.1007/s11060-004-8093-6. PMID 16215811
- [Background] Patchell RA, Tibbs PA, Regine WF, Dempsey RJ, Mohiuddin M, Kryscio RJ, Markesbery WR, Foon KA, Young B. Postoperative radiotherapy in the treatment of single metastases to the brain: a randomized trial. JAMA. 1998 Nov 4;280(17):1485-9. doi: 10.1001/jama.280.17.1485. PMID 9809728
- [Background] Roman DD, Sperduto PW. Neuropsychological effects of cranial radiation: current knowledge and future directions. Int J Radiat Oncol Biol Phys. 1995 Feb 15;31(4):983-98. doi: 10.1016/0360-3016(94)00550-8. PMID 7860415
- [Background] DeAngelis LM, Delattre JY, Posner JB. Radiation-induced dementia in patients cured of brain metastases. Neurology. 1989 Jun;39(6):789-96. doi: 10.1212/wnl.39.6.789. PMID 2725874
- [Background] Chang EL, Wefel JS, Maor MH, Hassenbusch SJ 3rd, Mahajan A, Lang FF, Woo SY, Mathews LA, Allen PK, Shiu AS, Meyers CA. A pilot study of neurocognitive function in patients with one to three new brain metastases initially treated with stereotactic radiosurgery alone. Neurosurgery. 2007 Feb;60(2):277-83; discussion 283-4. doi: 10.1227/01.NEU.0000249272.64439.B1. PMID 17290178
- [Background] Welzel G, Fleckenstein K, Schaefer J, Hermann B, Kraus-Tiefenbacher U, Mai SK, Wenz F. Memory function before and after whole brain radiotherapy in patients with and without brain metastases. Int J Radiat Oncol Biol Phys. 2008 Dec 1;72(5):1311-8. doi: 10.1016/j.ijrobp.2008.03.009. Epub 2008 Apr 28. PMID 18448270
- [Background] Li J, Bentzen SM, Li J, Renschler M, Mehta MP. Relationship between neurocognitive function and quality of life after whole-brain radiotherapy in patients with brain metastasis. Int J Radiat Oncol Biol Phys. 2008 May 1;71(1):64-70. doi: 10.1016/j.ijrobp.2007.09.059. PMID 18406884
- [Background] Masterton RA, Carney PW, Jackson GD. Cortical and thalamic resting-state functional connectivity is altered in childhood absence epilepsy. Epilepsy Res. 2012 May;99(3):327-34. doi: 10.1016/j.eplepsyres.2011.12.014. Epub 2012 Jan 24. PMID 22281064
- [Background] Sawrie SM, Chelune GJ, Naugle RI, Luders HO. Empirical methods for assessing meaningful neuropsychological change following epilepsy surgery. J Int Neuropsychol Soc. 1996 Nov;2(6):556-64. doi: 10.1017/s1355617700001739. PMID 9375160
- [Background] Kriegeskorte N, Simmons WK, Bellgowan PS, Baker CI. Circular analysis in systems neuroscience: the dangers of double dipping. Nat Neurosci. 2009 May;12(5):535-40. doi: 10.1038/nn.2303. PMID 19396166
- [Background] Luna B, Velanova K, Geier CF. Methodological approaches in developmental neuroimaging studies. Hum Brain Mapp. 2010 Jun;31(6):863-71. doi: 10.1002/hbm.21073. PMID 20496377
- [Background] Viviani R. Unbiased ROI selection in neuroimaging studies of individual differences. Neuroimage. 2010 Mar;50(1):184-9. doi: 10.1016/j.neuroimage.2009.10.085. Epub 2009 Nov 6. PMID 19900563
- [Background] Lie CH, Specht K, Marshall JC, Fink GR. Using fMRI to decompose the neural processes underlying the Wisconsin Card Sorting Test. Neuroimage. 2006 Apr 15;30(3):1038-49. doi: 10.1016/j.neuroimage.2005.10.031. Epub 2006 Jan 18. PMID 16414280
- [Background] Bhatnagar AK, Flickinger JC, Kondziolka D, Lunsford LD. Stereotactic radiosurgery for four or more intracranial metastases. Int J Radiat Oncol Biol Phys. 2006 Mar 1;64(3):898-903. doi: 10.1016/j.ijrobp.2005.08.035. Epub 2005 Dec 9. PMID 16338097
- [Background] Bhatnagar AK, Kondziolka D, Lunsford LD, Flickinger JC. Recursive partitioning analysis of prognostic factors for patients with four or more intracranial metastases treated with radiosurgery. Technol Cancer Res Treat. 2007 Jun;6(3):153-60. doi: 10.1177/153303460700600301. PMID 17535022